CLINICAL TRIAL: NCT00266201
Title: Evaluation of Biochemical Markers of Neurohumoral Activity and Correlation With Clinically Significant Parameters in Patients With Right Ventricular Failure and Congenital Heart Defects
Brief Title: Right Ventricular Failure in Congenital Heart Defects
Status: Completed | Type: Observational
Sponsor: Competence Network for Congenital Heart Defects (Other Government)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Other Study IDs: MP 5.1; 01G10210
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2007-04

CONDITIONS: Heart Failure; Congenital Heart Defects
Keywords: Heart Defects, Congenital; Right Ventricular Dysfunction; Low Cardiac Output; Biochemical markers; Neurohumoral activity
MeSH Terms: conditions — Heart Failure; Heart Defects, Congenital; Ventricular Dysfunction, Right; Cardiac Output, Low

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Usually, "heart failure" refers to myocardial insufficiency of the left ventricle. However, in patients with congenital heart defects, often predominantly the right ventricle is affected.

Brain natriuretic peptide (BNP) has been shown to be a reliable biomarker for left ventricular function and severity of left ventricular failure.

The objective of the present investigation is to evaluate brain natriuretic peptide (BNP) with regard to its predictive value as a biomarker for right ventricular function, clinical symptoms and/or the patients' quality of life.To this end, blood levels of neurohumoral markers are measured and tested for statistical correlation with exercise tolerance and right ventricular function, as assessed by imaging methods. A sample of healthy volunteers serves as a control group.

DETAILED DESCRIPTION:
Usually, "heart failure" refers to myocardial insufficiency of the left ventricle. In patients with congenital heart defects, predominantly the right ventricle and secondarily the right atrium and the pulmonary vasculature are affected. Due to advancing treatment options and the resulting higher life expectancy of patients with congenital heart defects, the number of these patients is increasing steadily. As, for these patients, right ventricular failure often is the factor limiting quality of life and life-span, evidence based drug treatment is both clinically important and of relevance with respect to health policy and health economics.

Concerning left ventricular failure, large controlled and randomised studies in the past years have provided evidence that treatment with beta-adrenergic blockers improves the systolic left ventricular function and decreases mortality in cases of left ventricular failure. These therapeutic achievements corroborated the hypothesis that stimulation of the neurohumoral, particularly the noradrenergic, system is a pathophysiological mechanism significant for the development of left ventricular failure.

Large studies demonstrated that brain natriuretic peptide (BNP) is a sensitive biomarker for activation of the noradrenergic system. Plasma levels of BNP closely correlate with the severity of left ventricular failure, qualifying BNP also as a marker of success/failure of treatment.

If right ventricular dysfunction also involves stimulation of the neurohumoral axis, it is conceivable that BNP in this condition also is a sensitive biomarker for activation of the noradregergic system. Under this condition BNP levels might also serve as a predictive marker for clinical outcome and success/failure of therapy as well.

The objective of the present investigation is to assess the predictive value of BNP as a biomarker for right ventricular function, clinical symptoms and/or the patients' quality of life. For this purpose, blood levels of neurohumoral markers are measured and tested for statistical correlation with exercise tolerance and right ventricular function, as assessed by imaging methods. A sample of healthy volunteers serves as a control group.

ELIGIBILITY:
Inclusion Criteria:

Patient group:

* Adolescents (at least14 years old)/adults with a surgically treated congenital heart defect that leads to stress of the right ventricle
* Consent of the patient, in the case of minors additional consent of the parents or the legal representative, to participation in the study.

Control group:

* Healthy population, comparable to the patient sample with respect to age and gender
* No heart defect, normal echocardiogram, ECG and MRI
* Consent of the test person, in case of minors additional consent of the parents or the legal representative, to participation

Exclusion Criteria

* Other clinically significant illnesses (e.g. malignant disease, impaired thyroid function)
* Morphological right ventricle as systemic ventricle
* Haemodynamically relevant left ventricular failure
* Treatment with a beta blocker

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient group:
  - Adolescents (at least14 years old)/adults with a surgically treated congenital heart
  Control group:
  - Healthy population, comparable to the patient sample with respect to age and gender
Sampling Method: Non-Probability Sample
Enrollment: 150
Dates: Start 2003-06; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Stiller, MD, Principal Investigator — German Heart Institute
Locations (9):
- Germany (9):
  - Zentrum fuer Kinderheilkunde und Jugendmedizin, Freiburg im Breisgau, Baden-Wurttemberg
  - Kinderherzzentrum des Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Herzzentrum Hamburg, UKE, Hamburg, Hamburg
  - Städtische Kliniken Oldenburg, Oldenburg, Lower Saxony
  - Herz- und Diabeteszentrum, Bad Oeynhausen, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Deutsches Kinderherzzentrum, Sankt Augustin, North Rhine-Westphalia
  - Deutsches Herzzentrum Berlin, Berlin, State of Berlin

REFERENCES:
- [Derived] Lemmer J, Heise G, Rentzsch A, Boettler P, Kuehne T, Dubowy KO, Peters B, Lemmer B, Hager A, Stiller B; German Competence Network for Congenital Heart Defects. Right ventricular function in grown-up patients after correction of congenital right heart disease. Clin Res Cardiol. 2011 Apr;100(4):289-96. doi: 10.1007/s00392-010-0241-8. Epub 2010 Oct 28. PMID 20981430